CLINICAL TRIAL: NCT00349947
Title: Abdominal Aortic Aneurysms: Simple Treatment or Prevention (AAA: STOP)
Brief Title: Exercise Therapy to Treat Adults With Abdominal Aortic Aneurysms
Acronym: AAA:STOP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 391; 5P50HL083800 (NIH); P50HL083800-01 (NIH)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will take part in an exercise program.
  Interventions: Behavioral: Exercise Program
- 2 (No Intervention): Participants will take part in a usual activity group.

INTERVENTIONS:
Behavioral: Exercise Program — Participants who live within 15 miles of the Palo Alto VA Hospital will take part in a supervised aerobic exercise program 3 days a week. Participants who live farther than 15 miles from the hospital will receive a detailed exercise plan and will exercise on their own while wearing a heart rate and activity tracking device. They will also attend monthly study visits for review of their progress. All participants assigned to the exercise program will be encouraged to increase their daily exercise. Each day they will wear a pedometer; twice a month they will wear a global positioning system (GPS) and heart rate monitor.
  Arms: 1

SUMMARY:
An abdominal aortic aneurysm (AAA) is a weakened and enlarged area in the abdominal aorta, which is a large blood vessel in the abdomen. If an AAA ruptures, it can be life-threatening. Research has shown that sedentary individuals are at increased risk of developing AAAs. This study will evaluate the effectiveness of an exercise program at limiting the growth of small AAAs in older individuals.

DETAILED DESCRIPTION:
AAAs are common among older individuals, and are the 10th leading cause of death for men over the age of 55. A ruptured AAA usually leads to death. Therefore, early detection and treatment are critical. Currently, there are several surgical treatment options available, but there is no proven non-surgical treatment for AAAs. Research has shown that physical inactivity may be linked to the development of AAAs. The purpose of this study is to gather information on AAA risk factors, and to evaluate the effectiveness of an exercise program at preventing the growth of small AAAs in older individuals.

This study will be composed of three individual projects. Project 1 will enroll 1400 individuals with small AAAs. Project 2 will enroll 1000 individuals with unknown aortic size and previously tested exercise capacity. Both groups of participants will attend one study visit, at which time their medical history and physical activity history will be recorded, vital signs will be collected, and blood and urine sample will be given. Questionnaires will be completed to document physical activity levels and AAA risk factors. An abdominal ultrasound will be performed to measure the size of the aorta or AAA. Participants in Project 2 will also take part in a treadmill exercise test, during which heart rate and blood pressure will be recorded, and heart activity will be monitored by an electrocardiogram (ECG).

The third project will last 3 years and will enroll 340 individuals from Project 1. Participants will be randomly assigned to either an exercise program or a usual activity group. An initial screening visit will include medical history review, vital sign measurements, blood collection, questionnaires, an abdominal ultrasound, a positron emission tomography (PET) scan, a computed tomography (CT) scan, and a magnetic resonance imaging (MRI) scan.

Participants in the exercise program will complete an exercise test at the beginning of the study and every 6 months for the duration of the study. Participants who live within 15 miles of the Palo Alto VA Hospital will take part in a supervised aerobic exercise program 3 days a week. Participants who live farther than 15 miles from the hospital will receive a detailed exercise plan and will exercise on their own while wearing a heart rate and activity tracking device. They will also attend monthly study visits for review of their progress. All participants assigned to the exercise program will be encouraged to increase their daily exercise. Each day they will wear a pedometer; twice a month they will wear a global positioning system (GPS) and heart rate monitor. Participants assigned to the usual activity group will wear pedometers each day and will maintain their usual level of physical activity. At yearly study visits, blood will be collected and physical activity levels will be assessed.

All Project 3 participants with AAAs smaller than 4 cm will undergo an ultrasound and blood collection once a year; participants with AAAs 4 cm or larger will undergo the same procedures every 6 months. At the end of 3 years, all participants will attend a final study visit at which time their medical history will be reviewed and blood will be collected. They will also undergo an abdominal ultrasound, and PET, CT, and MRI scans.

ELIGIBILITY:
Inclusion Criteria:

* Small AAA less than 5.5 cm in size
* Over age 50

Exclusion Criteria:

* Patients with congenital aneurysm syndromes such as Ehlers-Danlos' or Marfan's

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2006-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Growth rate of AAAs | Measured at Year 3

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L. Dalman, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Palo Alto Veterans Affairs Health Care System, Palo Alto, California
  - Kaiser Permanente Hospitals of Northern California, Santa Clara, California
  - Stanford University Medical Center, Stanford, California

REFERENCES:
- [Derived] Vainshelboim B, Rao S, Chan K, Lima RM, Ashley EA, Myers J. A comparison of methods for determining the ventilatory threshold: implications for surgical risk stratification. Can J Anaesth. 2017 Jun;64(6):634-642. doi: 10.1007/s12630-017-0862-8. Epub 2017 Apr 5. PMID 28382529
- [Derived] Bianchi VE, Herbert WG, Myers J, Ribisl PM, Miller LE, Dalman RL. Relationship of obstructive sleep apnea and cardiometabolic risk factors in elderly patients with abdominal aortic aneurysm. Sleep Breath. 2015 May;19(2):593-8. doi: 10.1007/s11325-014-1053-2. Epub 2014 Sep 10. PMID 25204854
- [Derived] Betz HH, Myers J, Jaffe A, Smith K, Dalman R. Reproducibility of the Veterans Physical Activity Questionnaire in an elderly population. J Phys Act Health. 2015 Mar;12(3):376-81. doi: 10.1123/jpah.2013-0124. Epub 2014 Apr 17. PMID 24763187
- [Derived] Myers J, McElrath M, Jaffe A, Smith K, Fonda H, Vu A, Hill B, Dalman R. A randomized trial of exercise training in abdominal aortic aneurysm disease. Med Sci Sports Exerc. 2014 Jan;46(1):2-9. doi: 10.1249/MSS.0b013e3182a088b8. PMID 23793234
- [Derived] Myers J, Dupain M, Vu A, Jaffe A, Smith K, Fonda H, Dalman R. Agreement between activity-monitoring devices during home rehabilitation: a substudy of the AAA STOP trial. J Aging Phys Act. 2014 Jan;22(1):87-95. doi: 10.1123/japa.2012-0133. Epub 2013 Feb 14. PMID 23416349